CLINICAL TRIAL: NCT04737083
Title: Evaluation of CGH Array in Prenatal Diagnosis of Bilateral Clubfoot
Brief Title: CGH Array in Bilateral Clubfoot
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Matthieu DAP, medical doctor (MD), Central Hospital, Nancy, France
Other Study IDs: 2021PI006
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-01

CONDITIONS: Clubfoot; Prenatal Disorder
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- clubfoot fetuses
  Interventions: Genetic: CGH array

INTERVENTIONS:
Genetic: CGH array — a CGH array is systematically offer to women when the fetus show bilateral clubfoot during prenatal ultrasound screening

SUMMARY:
In prenatal diagnosis of isolated bilateral clubfoot our team propose genetic analysis: a CGH-array. We want to study the rate of aberrations in these cases.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* fetus with isolated bilateral clubfoot

Exclusion Criteria:

* no

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Study Population: Pregnant women who had their follow-up in our team with a prenatal diagnosis of bilateral clubfoot in their fetus.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
rate of abnormal CGH-array in the population | 9 months

SECONDARY OUTCOMES:
type of abnormalities in CGH-array study | 9 months